CLINICAL TRIAL: NCT03689231
Title: Volumetric Imaging Follow up of Patients With Liver Metastases of Small Intestinal Neuroendocrine Tumors (NETs).
Acronym: VOLUNET
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: VOLUNET
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Neuroendocrine Tumors; Liver Metastases
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Volumetric measurements of liver metastases — Depending on the available data and to be reproducible, patients will be divided into 2 sub-groups of follow-up imaging: CT only or MRI only, combined evaluation being not reliable for tumor detection
  Patient follow-up at CT or MRI will be analyzed at baseline (date of discovery of hepatic metastatic disease), then 3-6 months after the start of the study, then annually.
  At each assessment, a radiologist will analyze: the total volume of liver metastases (mm3), the estimated volume of the two target lesions chosen for RECIST follow-up (mm3), the number of liver lesions, and the evolution according to the RECIST criteria based on uni-dimensional measurements.
  We will then correlate the following clinical data collected for patients: age, sex, presence of a carcinoid syndrome, Ki67 (%) and chromogranin A blood level (%) at diagnosis, number and location of other metastases, Octreoscan or Stereotactic Radio Surgery data if available.

SUMMARY:
More than 50% of intestinal NETs are metastatic at the time of diagnosis, the liver being the main affected organ in 50-90% of cases.

Initial liver tumor burden and slope of the tumor growth rate are two major prognostic factors in patients with intestinal NETs, followed by tumor grade at pathology. They are used in routine practice by oncologists to adapt patient treatment.

Unlike other tumors, most NETs metastases are slow-growing tumors. Previous studies have shown that approximately half of the patients diagnosed with liver metastases showed no progression over a period of 3 to 6 months.

The aim of this non randomised retrospective cohort study is to investigate whether the volumetric monitoring of the total tumor burden compared to the RECIST 1.1 criteria (used in routine practice by radiologists) at baseline and early follow-up (3 to 6 months) is more suitable for NETs, making possible to predict the prognosis at the onset of the disease, and also allowing a better adaptation of the treatment.

The secondary objectives are to evaluate if the initial volume of the liver tumor is a prognostic factor of time to progression, to correlate the initial liver tumor volume and the number of liver lesions to the blood concentration of Chromogranin A (CgA), the presence of extra-abdominal disease and to correlate the tumor growth rate (TGR) and KI 67 (%) at base-line.

ELIGIBILITY:
Inclusion Criteria:

* Well differentiated intestinal neuroendocrine tumor with at least one liver metastasis
* The liver metastasis must be visible and measurable on CT scans or MRI
* Patients monitored without invasive liver treatment : surgery, RF ablation / Trans-arterial chemoembolization
* Patients monitored without systemic treatment such as: Chemotherapy, Everolimus, Sunitinib (Somatostatin analogues allowed)
* Surgery of the primary tumor allowed

Exclusion Criteria:

* Other type of NETs
* Absence of liver metastases
* Liver metastases not visible on CT scans/MRI, poorly limited lesions and small target lesions ( less than 10mm) that are difficult to measure
* Lesions visible only on diffusion-weighted imaging -MRI acquisitions, thus presenting poorly limited contours
* Invasive liver treatment : surgery, Radio frequency / Trans-arterial chemoembolization
* Systemic treatments: Chemotherapy / Everolimus / Sunitinib
* Insufficient follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old, with intestinal well differentiated intestinal neuroendocrine tumor and with at least one liver metastasis, without any invasive or systemic treatment for liver metastasis (Somatostatin analogues only allowed).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Could the evolution of the initial liver tumor volume (on two follow-up CT scans / MRI over a period of 3 to 6 months) be predictive of progression-free survival according to the RECIST criteria? | 6 months
  To assess if the evolution of the initial liver tumor volume compared to a follow-up CT scans / MRI over a period of 3 to 6 months is predictive of progression-free survival according to the RECIST criteria

SECONDARY OUTCOMES:
Could the evolution of the initial liver tumor volume (on two follow-up CT scans / MRI over a period of 3 to 6 months) be predictive of progression-free survival according to the RECIST criteria? | 6 months
  To evaluate whether the initial volume of the liver tumor is a prognostic factor of time to progression
Could the evolution of the initial liver tumor volume (on two follow-up CT scans / MRI over a period of 3 to 6 months) be predictive of progression-free survival according to the RECIST criteria? | 6 months
  To determine the tumor growth rate
Could the evolution of the initial liver tumor volume (on two follow-up CT scans / MRI over a period of 3 to 6 months) be predictive of progression-free survival according to the RECIST criteria? | 6 months
  To estimate the evolution of tumor volume as a function of time that may anticipate earlier than RECIST the tumor growth
Could the evolution of the initial liver tumor volume (on two follow-up CT scans / MRI over a period of 3 to 6 months) be predictive of progression-free survival according to the RECIST criteria? | 6 months
  To correlate the initial liver tumor volume and the number of liver lesions to the blood concentration of Chromogranin A (CgA) and the presence of extra-abdominal disease.
Could the evolution of the initial liver tumor volume (on two follow-up CT scans / MRI over a period of 3 to 6 months) be predictive of progression-free survival according to the RECIST criteria? | 6 months
  To correlate the tumor growth rate (TGR) and KI 67 (%) at base-line (on liver metastasis if available or on primary tumor)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de radiologie-Pavillon B-Cellule Recherche imagerie - Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No